CLINICAL TRIAL: NCT06378879
Title: Intermittent Boluses Versus Continuous Infusion of Propofol During Standard Upper Endoscopy
Brief Title: Intermittent Boluses Versus Infusion of Propofol During Gastroscopy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Balqa Applied University (Other)
Collaborators: Luzmila Hospital (Unknown)
Responsible Party: Principal Investigator, Tarek Mazzawi, Assistant Professor, Al-Balqa Applied University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 1073/1/3/26
Record Dates: First submitted 2024-03-30; First posted 2024-04-23 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Anesthesia
Keywords: Propofol; Dormicum; Infusion; Bolus; Gastroscopy
MeSH Terms: interventions — Propofol; Injections

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Continuous infusion (CI group) of propofol (Active Comparator): CI was defined by continuous propofol infusion at a 3 mg/ kg/h rate with induction using benzodiazepine (2 mg dormicum i.v.) to evaluate the effect of the drug and assess sedation induction time, total dose of propofol, recovery time, quality of sedation.
  Interventions: Drug: Propofol 100 MG in 10 ML Injection
- Intermittent bolus injection (BI group) of propofol (Active Comparator): BI was defined by intermittent use of 20 mg propofol boluses on demand, with a minimum period of 30 seconds between boluses to evaluate the effect of the drug and assess sedation induction time, total dose of propofol, recovery time, quality of sedation.
  Interventions: Drug: Propofol 100 MG in 10 ML Injection

INTERVENTIONS:
Drug: Propofol 100 MG in 10 ML Injection — Sedation induction time (minutes), total dose of propofol (mg), recovery time (minutes), any involuntary patient movement, quality of sedation (VAS) and adverse events
  Other Names: Diprivan (100mg/10ml)

SUMMARY:
It is unclear whether continuous infusion or intermittent bolus injection of propofol is better for achieving adequate sedation during a standard upper endoscopy. The study aimed to compare the efficacy and safety of continuous infusion and intermittent bolus injection of Propofol (Diprivan) during a standard upper endoscopy. In this prospective study, patients will be randomly assigned to undergo a standard upper endoscopy with either continuous infusion (CI group) or intermittent bolus injection (BI group) of Propofol (Diprivan) administered by an anesthesiologist. The primary outcome will be to assess the quality of sedation by the endoscopist (VAS). In addition to other sedation-related parameters that will include sedation induction time (minutes), total dose of propofol (mg), recovery time (minutes) using Aldrete score, any involuntary patient movement, and adverse events.

DETAILED DESCRIPTION:
Patients of both genders, aged between 18 and 85 years old and referred to standard upper endoscopy at Luzmila Hospital will be included in the study. Patients who are pregnant, have known allergies to the drugs used or a history of sedation-related complications (i.e., severe paradoxical response, hypoxemia, bradycardia, and hypotension) or gastrectomy, are American Society of Anesthesiologist (ASA) class ≥ IV (11), or are unable to provide informed consent will be excluded from participating in the study. The patients undergoing a standard upper endoscopy will be randomly assigned to either continuous infusion (CI group) of propofol (Diprivan) with induction using benzodiazepine (2 mg Dormicum i.v.) or only intermittent bolus injection (BI group) of propofol (Diprivan) infused by an anesthesiologist. BI was defined by intermittent use of 20 mg propofol (Diprivan) boluses on demand, with a minimum period of 30 seconds between boluses to evaluate the effect of the drug. CI was defined by continuous propofol (Diprivan) infusion at a 3 mg/ kg/h rate.

The anesthesiologist will follow up the patient during the first observation period, the average time spent in the recovery area and register the requied data during the procedure using Aldrete score (a post anesthesia recovery score where a minimum score of 8 is required for discharge).

The patients' identities will be coded and the data will be kept confidential. The study protocol will be performed according to the Decalrations of Helsinki and will be applied for approval by the Institutional Review Board at Al-Balqa Applied University. Written informed consent was obtained from all patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both genders
* Age between 18 and 85 years old
* Referred to standard upper endoscopy at Luzmila Hospital

Exclusion Criteria:

* Patients who are pregnant,
* Known allergies to the used drugs
* History of sedation-related complications (i.e., severe paradoxical response, hypoxemia, bradycardia, and hypotension)
* Previous history of gastrectomy,
* Patients are American Society of Anesthesiologist (ASA) class ≥ IV ,
* Patients are unable to provide informed consent

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-09-06 (Estimated); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-07-30 (Estimated)

PRIMARY OUTCOMES:
Sedation induction time (minutes) | 30 minutes
  Sedation induction time (minutes) is the time measured from the deep sedation induction until the patient is deeply sedated
Total dose of propofol (mg) | 30 minutes
  Total dose of propofol (mg) used during the upper endoscopy procedure
Recovery time (minutes) | 30 minutes
  Recovery time (minutes) is the time used for the patients to open their eyes after stoping sedation

SECONDARY OUTCOMES:
Involuntary movement | 30 minutes
  Any involuntary patient movement during the endoscopy procedure under deep sedation
Quality of sedation | 30 minutes
  How deeply is the patient sedated (VAS) as assessed by the endoscopist (1 good, 2 moderate, 3 poor)
Adverse events | 30 minutes
  Any adverse events occurring during the procedure such as apnea, dyspnea, hiccups, jerky movements...etc

CONTACTS AND LOCATIONS:
Overall Officials: Tarek Mazzawi, MD, PhD, Principal Investigator — Faculty of Medicine, Al-Balqa Applied University

IPD SHARING:
Plan to Share IPD: Yes
The analysis and results will be published in peer-reviewed journal. Study protocol, statistical analysis plan, informed consent will be provided upon request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: During 2025
Access Criteria: According to publishing journal

REFERENCES:
- [Background] Gonzalez-Santiago JM, Martin-Noguerol E, Vinagre-Rodriguez G, Hernandez-Alonso M, Duenas-Sadornil C, Perez-Gallardo B, Mateos-Rodriguez JM, Fernandez-Bermejo M, Robledo-Andres P, Molina-Infante J. Intermittent boluses versus pump continuous infusion for endoscopist-directed propofol administration in colonoscopy. Rev Esp Enferm Dig. 2013 Aug;105(7):378-84. doi: 10.4321/s1130-01082013000700002. PMID 24206547
- [Background] Cohen LB, Wecsler JS, Gaetano JN, Benson AA, Miller KM, Durkalski V, Aisenberg J. Endoscopic sedation in the United States: results from a nationwide survey. Am J Gastroenterol. 2006 May;101(5):967-74. doi: 10.1111/j.1572-0241.2006.00500.x. PMID 16573781
- [Background] Jung M, Hofmann C, Kiesslich R, Brackertz A. Improved sedation in diagnostic and therapeutic ERCP: propofol is an alternative to midazolam. Endoscopy. 2000 Mar;32(3):233-8. doi: 10.1055/s-2000-96. PMID 10718389
- [Background] Riphaus A, Stergiou N, Wehrmann T. Sedation with propofol for routine ERCP in high-risk octogenarians: a randomized, controlled study. Am J Gastroenterol. 2005 Sep;100(9):1957-63. doi: 10.1111/j.1572-0241.2005.41672.x. PMID 16128939
- [Background] McQuaid KR, Laine L. A systematic review and meta-analysis of randomized, controlled trials of moderate sedation for routine endoscopic procedures. Gastrointest Endosc. 2008 May;67(6):910-23. doi: 10.1016/j.gie.2007.12.046. PMID 18440381
- [Background] Dumonceau JM, Riphaus A, Aparicio JR, Beilenhoff U, Knape JT, Ortmann M, Paspatis G, Ponsioen CY, Racz I, Schreiber F, Vilmann P, Wehrmann T, Wientjes C, Walder B; NAAP Task Force Members. European Society of Gastrointestinal Endoscopy, European Society of Gastroenterology and Endoscopy Nurses and Associates, and the European Society of Anaesthesiology Guideline: Non-anesthesiologist administration of propofol for GI endoscopy. Endoscopy. 2010 Nov;42(11):960-74. doi: 10.1055/s-0030-1255728. Epub 2010 Nov 11. PMID 21072716
- [Background] ASGE Standards of Practice Committee; Early DS, Lightdale JR, Vargo JJ 2nd, Acosta RD, Chandrasekhara V, Chathadi KV, Evans JA, Fisher DA, Fonkalsrud L, Hwang JH, Khashab MA, Muthusamy VR, Pasha SF, Saltzman JR, Shergill AK, Cash BD, DeWitt JM. Guidelines for sedation and anesthesia in GI endoscopy. Gastrointest Endosc. 2018 Feb;87(2):327-337. doi: 10.1016/j.gie.2017.07.018. Epub 2018 Jan 3. No abstract available. PMID 29306520
- [Background] Riphaus A, Geist C, Schrader K, Martchenko K, Wehrmann T. Intermittent manually controlled versus continuous infusion of propofol for deep sedation during interventional endoscopy: a prospective randomized trial. Scand J Gastroenterol. 2012 Sep;47(8-9):1078-85. doi: 10.3109/00365521.2012.685758. Epub 2012 May 28. PMID 22631051
- [Background] Hendrix JM, Garmon EH. American Society of Anesthesiologists Physical Status Classification System. 2025 Feb 11. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK441940/ PMID 28722969
- [Background] Roelandt P, Haesaerts R, Demedts I, Bisschops R. Implementation of the Aldrete score reduces recovery time after non-anesthesiologist-administered procedural sedation in gastrointestinal endoscopy. Endosc Int Open. 2022 Dec 15;10(12):E1544-E1547. doi: 10.1055/a-1964-7458. eCollection 2022 Dec. PMID 36531676
- See also: University website — http://www.bau.edu.jo